CLINICAL TRIAL: NCT00313170
Title: Phase II Study to Evaluate the Efficacy and Tolerability of Fulvestrant 250mg, 250mg Plus 250mg Loading Regimen and 500mg in Postmenopausal Women With ER +ve Advanced Breast Cancer Progressing or Relapsing After Previous Endocrine Therapy
Brief Title: A Clinical Trial to Compare Efficacy and Tolerability of Fulvestrant 250mg, 250mg Plus 250mg Loading Regimen and 500mg
Acronym: FINDER II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6997C00006; FINDER II
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: oncology; cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Fulvestrant 250 mg (intramuscular injection 250 mg)
  Interventions: Drug: Fulvestrant
- 2 (Experimental): Fulvestrant 250 mg (+ 250 mg loading regimen)
  Interventions: Drug: Fulvestrant
- 3 (Experimental): Fulvestrant 500 mg (intramuscular injection 500 mg)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection 250 mg & 500 mg
  Other Names: Faslodex; ZD9238

SUMMARY:
This study will assess the relationship between fulvestrant dose and efficacy in postmenopausal women with oestrogen receptor positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer has continued to grow after having received treatment with an anti-estrogen hormonal treatment such as tamoxifen or an aromatase inhibitor.
* Requiring hormonal treatment.
* Postmenopausal women (woman who has stopped having menstrual periods)

Exclusion Criteria:

* Treatment with more than one previous regimen of systemic anticancer therapy other than endocrine therapy for advanced BC.
* Treatment with more than one previous regimen of endocrine therapy for advanced BC.
* An existing condition that prevents compliance.

Ages: 45 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-05-30 (Actual); Primary Completion 2008-06-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Breast Cancer Established Brands Team Medical Science Director, MD, Study Director — AstraZeneca
Locations (32):
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Wilrijk
- Canada (9):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, London, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (3):
  - Research Site, Cheb
  - Research Site, Jičín
  - Research Site, Prague
- France (4):
  - Research Site, Bordeaux
  - Research Site, Brivé
  - Research Site, Clermont-Ferrand
  - Research Site, Poitiers
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Szeged
  - Research Site, Tatabánya
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Olsztyn
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Research Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Pritchard KI, Rolski J, Papai Z, Mauriac L, Cardoso F, Chang J, Panasci L, Ianuli C, Kahan Z, Fukase K, Lindemann JP, Macpherson MP, Neven P. Results of a phase II study comparing three dosing regimens of fulvestrant in postmenopausal women with advanced breast cancer (FINDER2). Breast Cancer Res Treat. 2010 Sep;123(2):453-61. doi: 10.1007/s10549-010-1022-9. Epub 2010 Jul 15. PMID 20632084
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=407&filename=CSR-D6997C00006.pdf
- See also: CSR-D6997C00006.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=407&filename=CSR-D6997C00006.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with oestrogen receptor positive advanced breast cancer progressing or relapsing after previous endocrine therapy were randomised between 30th May 2006 and 30th November 2007
Groups:
- Fulvestrant 250 mg: Fulvestrant 250 mg
- Fulvestrant 250 mg + Loading Dose: Fulvestrant 250 mg + Loading Dose
- Fulvestrant 500 mg: Fulvestrant 500 mg
Period: Overall Study
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Started | 47 | 51 | 46
Completed | 11 | 17 | 14
Not Completed | 36 | 34 | 32
Not completed — Death | 2 | 4 | 2
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Disease progression | 31 | 26 | 27
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Incorrect enrollment | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Progression (investigators opinion) | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg | Total
Number analyzed (Participants) | 47 | 51 | 46 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.9) | 68.1 (9.9) | 65.5 (9.0) | 65.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 46 | 144
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 45 | 51 | 46 | 142
  Oriental (Japanese) | 1 | 0 | 0 | 1
  Oriental (Asian other than Chinese or Japanese) | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (ORR)
Description: Objective response rate was defined as percentage of patients with either complete response (CR - disappearance of all target lesions) or partial response (PR - at least 30% decrease in the sum of diameters of target lesions). All patients were to be followed up every 12 weeks for progression, defined by response evaluation criteria in solid tumors (RECIST v1.1).
Time Frame: The planned data cut-off for this study was when all patients, except withdrawals, had been followed up for at least 24 weeks. Patients received treatment up to approximately 2 years.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 47 | 51 | 46
Percentage of patients | 8.5 [2.4 to 20.4] | 5.9 [1.2 to 16.2] | 15.2 [6.3 to 28.9]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time from randomisation until objective disease progression or death (in the absence of objective progression) using the Kaplan-Meier method. RECIST tumor assessments were carried out every 12 weeks until progression.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 47 | 51 | 46
Days | 88 [79 to 260] | 172 [80 to 339] | 169 [82 to 477]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from date of first documentation of the response (CR or PR) until the date of disease progression or death from any cause.
Time Frame: as for outcome 1
Population: All objective responders
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 4 | 3 | 7
Days | NA [NA to NA] — not estimable | NA [66 to NA] — median and 75th percentile not estimable | 539 [539 to 539]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the proportion of all randomised patients who had clinical benefit (response of CR, PR or SD>=24 weeks.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 47 | 51 | 46
Percentage of patients | 31.9 [19.1 to 47.1] | 47.1 [32.9 to 61.5] | 47.8 [32.9 to 63.1]

5. Secondary Outcome: Pharmacokinetic Parameter: Mean Population Clearance, a Measure of the Efficiency With Which Fulvestrant is Eliminated From the Body
Description: A 2-compartment model with a 1st order absorption and 1st order elimination process was fitted to the fulvestrant concentration-time data. Relative standard error is reported for the mean.
Time Frame: Baseline to 12 weeks
Population: Participants who had PK samples only
Measure: Least Squares Mean (Standard Error); unit: litres per hour
Groups:
- Fulvestrant: Fulvestrant arms pooled
Arm/Group | Fulvestrant
Number analyzed (Participants) | 72
litres per hour | 31 (3.29)

6. Secondary Outcome: Pharmacokinetic Parameter: Mean Volume of Distribution at Steady State, a Measure of the Apparent Volume in the Body Into Which Fulvestrant Distributes
Description: A 2-compartment model with a 1st order absorption and 1st order elimination process was fitted to the fulvestrant concentration-time data. Relative standard error is reported for the mean. The mean estimate of volume of distribution at steady state was reported as the sum of V1/F and V2/F in the clinical study report.
Time Frame: Baseline to 12 weeks
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fulvestrant
Number analyzed (Participants) | 72
Liters
  V1/F | 20600 (3.67)
  V2/F | 35700 (27.8)

ADVERSE EVENTS:
Description: 1 patient in the 250mg + LD arm was randomised but did not receive any randomised therapy. This patient is included in the efficacy summaries but is excluded from the safety summaries.
  All-Cause Mortality: patients who died whilst on study treatment or during 56 days after the last fulvestrant injection.
  Serious Adverse Events: Patients with SAE other than death are reported.
  NOTE: Other Adverse Events include serious and non-serious AEs.
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
All-Cause Mortality (participants affected / at risk) | 2/47 | 4/50 | 2/46
Serious Adverse Events (participants affected / at risk) | 4/47 | 9/50 | 4/46
Other Adverse Events (participants affected / at risk) | 36/47 | 35/50 | 31/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=47) | Fulvestrant 250 mg + Loading Dose (N=50) | Fulvestrant 500 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Macular Hole (Eye disorders) | 1 | 0 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=47) | Fulvestrant 250 mg + Loading Dose (N=50) | Fulvestrant 500 mg (N=46)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 6
Nausea (Gastrointestinal disorders) | 12 | 9 | 7
Vomiting (Gastrointestinal disorders) | 3 | 4 | 5
Asthenia (General disorders) | 5 | 4 | 4
Fatigue (General disorders) | 4 | 11 | 7
Oedema Peripheral (General disorders) | 2 | 3 | 2
Injection Site Pain (General disorders) | 6 | 7 | 6
Herpes Zoster (Infections and infestations) | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 3 | 1
Weight Decreased (Investigations) | 1 | 6 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 0
Headache (Nervous system disorders) | 5 | 4 | 3
Anxiety (Psychiatric disorders) | 2 | 5 | 2
Depression (Psychiatric disorders) | 3 | 4 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Hot Flush (Vascular disorders) | 9 | 5 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less